CLINICAL TRIAL: NCT06692920
Title: Characterizing the Pathophysiological Role of the Pallido-thalamocortical Motor Pathway in Parkinson's Disease.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NEURO-2016-24971
Record Dates: First submitted 2024-11-13; First posted 2024-11-18 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Parkinson's patients with DBS surgery planned as part of routine clinical care
  Interventions: Other: DBS stimulation

INTERVENTIONS:
Other: DBS stimulation — * Standard of care DBS surgery
  * stimulation through the DBS lead during their DBS lead surgery, the study team will use 2 sets of stimulation settings on each participant:
    1. Stimulation through the DBS contact whose electrical activity is the MOST similar to the area of the brain that controls movement
    2. Stimulation through the DBS contact whose electrical activity is the LEAST similar to the area of the brain that controls movement

SUMMARY:
When a patient gets DBS surgery, the neurosurgeon makes a hole in the skull through which they can put the DBS lead down in deep parts of the brain that help control movement. For this study, research participants will also have an ECoG strip put through the same hole (no extra holes are being made for research purposes). The ECoG strip is a little less than half an inch wide, and a little more than 2.5 inches long. It is very, very thin; it is a thin plastic film with flat metal sensors that can record the electrical activity in the brain. The ECoG strips are FDA approved. The neurosurgeon will slide the ECoG strip under the skull but on top of the brain, over another area of the brain that helps control hand/arm movement (motor cortex), so that the study team can record the activity there. The study team will record brain activity from the DBS lead and the ECoG strip simultaneously to try to understand how the brain communicates and sends information. The study team will check that the ECoG strip is in the right place by delivering a very small electrical pulse to the wrist. If the ECoG strip is in the correct location, this electrical pulse will show up on the brain activity being recorded by the sensors in the ECoG strip. Fluoroscopy (i.e. X-ray images that can be taken quickly) will also be done at the end of the surgery to help confirm the location of the ECoG strip. During fluoroscopy, an X-ray beam is used to track a contrast agent ("X-ray dye") through the body, so that the body can be seen in detail. This involves some radiation exposure for the participant, so this is described in the consent form. Patients who want to sign up for the study will not be allowed to do so if they have had other radiation exposures within the past year that would go over a safe limit when added to the amount of radiation expected from the fluoroscopy for this study.

DETAILED DESCRIPTION:
The goal of this study is to understand the relationship between network brain activity and motor signs of Parkinson's disease, and to determine if brain activity can predict optimal locations or network pathways for stimulation. During deep brain stimulation lead placement surgery, research participants will have an FDA approved ECoG strip placed through the DBS lead burr hole over the primary motor cortex. The study team will record brain activity from the DBS lead and the ECoG strip simultaneously while the participant performs a reach-to-target motor task, to understand how different brain regions communicate and are associated with motor signs of Parkinson's disease. The study team will look for specific brain activity biomarkers hypothesized to be associated with Parkinson's disease and will then direct stimulation through the DBS lead toward regions showing those biomarkers and compare to stimulation directed to areas not showing the specified biomarkers. Neural pathways being activated by stimulation and behavioral measures of the reach task will be compared between the two stimulation conditions.

Intervention:

1. Stimulation through the DBS lead contact showing the most coherence with brain activity in the motor cortex
2. Stimulation through the DBS lead contact showing the least coherence with brain activity in the motor cortex

During the mapping session patients will either be asked to perform motor tasks such as finger-tapping, pronating/supinating the wrist, manipulating a joystick, or pointing to targets on a touch-sensitive, LCD positioned in front of them. Patients may also be asked to perform cognitive tasks such as maintaining items in working memory or deciding between potentially rewarding stimuli with either a joystick or a finger response pad.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD
* DBS surgery at UMN is planned as part of routine clinical care
* Aged 21-75

Exclusion Criteria:

* Other significant neurological disorder, which may confound neurophysiological changes associated with Parkinson's disease
* History of dementia
* Patients with post-operative complications or adverse effects (e.g. ON stimulation dystonias) that affect patient safety or confound the experiment will be excluded from further study
* Pregnant women
* Known research radiation exposure within the last year that is determined to be unsafe when compounded with the expected radiation dose from intraoperative fluoroscopy

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
amount of activity in the pallidothalamic pathway from stimulation, comparing the two sets of stimulation | post-surgery (1 day)
  The pallidothalamic pathway is what connects the two locations of the brain from which we are recording (GPi and motor cortex). We will also see how the two sets of stimulation made a difference in measurements of bradykinesia (slowness of movement): how long it took for the participant to get ready to move, how fast they started moving, and how long it took them to touch the startpad.
The relationship (slope) between the measures of bradykinesia and total pathway activation | post-surgery (1 day)
  will be estimated via a linear mixed-effects (LME) model that considers multiple subjects and multiple observations within subject

CONTACTS AND LOCATIONS:
Overall Officials: Joshua E Aman, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States